CLINICAL TRIAL: NCT06745882
Title: Prospective Trial to Assess Real-world Outcomes and Predictive Biomarkers of Response to Pembrolizumab With or Without Chemotherapy in Black Patients With NSCLC
Brief Title: Prospective Trial Assessing Real World Outcomes Response to Pembro in Black Patients w/ NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Foundation Medicine (Industry); Go-2 Lung (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21630
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Justice
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Carboplatin; Pemetrexed; pembrolizumab; Albumin-Bound Paclitaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Non-interventional prospective cohort and participants will receive standard of care pembrolizumab with or without chemotherapy.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Pembrolizumab; Drug: Abraxane; Drug: Paclitaxel
- Cohort 2: arm A (Experimental): Cohort 2 Arm A will enroll patients with NSCLC with PD-L1 TPS status ≥1% and ctDNA tumor fraction low/negative and be treated with pembrolizumab monotherapy.
  Interventions: Drug: Pembrolizumab
- Cohort 2: arm B (Experimental): Cohort 2 Arm B will enroll patients with NSCLC with any PD-L1 status and ctDNAtumor fraction intermediate/high -OR- PD-L1 TPS<1% and any ctDNA level treated with chemotherapy plus pembrolizumab.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Pembrolizumab; Drug: Abraxane; Drug: Paclitaxel

INTERVENTIONS:
Drug: Cisplatin — Given on day 1 of every 21-day cycle.
  Arms: Cohort 1; Cohort 2: arm B
Drug: Carboplatin — Given on day 1 of every 21-day cycle.
  Arms: Cohort 1; Cohort 2: arm B
Drug: Pemetrexed — Given on day 1 of every 21-day cycle.
  Arms: Cohort 1; Cohort 2: arm B
Drug: Pembrolizumab — Given on day 1 of every 21-day cycle. After cycle 4 is given every 6 weeks.
Drug: Abraxane — Given on days 1, 8, and 15 of each 21-day cycle.
  Arms: Cohort 1; Cohort 2: arm B
Drug: Paclitaxel — Given on day 1 of every 21-day cycle.
  Arms: Cohort 1; Cohort 2: arm B

SUMMARY:
This is a non-registrational, cohort study enrolling eligible Black patients diagnosed with histologically or cytologically, advanced/metastatic NSCLC without known EGFR/ALK/ROS1 tumor mutations, and who are ≥ 18 years of age, ECOG performance status 0-2, and may have detectable ctDNA at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent.
* Must be ≥ 18 years of age on day of signing informed consent.
* Be Black / African American per self-report.
* Have an ECOG performance status of 0- 2.
* Have histologically or cytologically confirmed, advanced/metastatic NSCLC.
* Be treatment naïve in the advanced/metastatic/recurrent disease setting.
* No known EGFR/ALK/ROS1 tumor mutations. Liquid biopsies are acceptable.
* Patients who received platinum-containing adjuvant chemotherapy, neoadjuvant chemotherapy or definitive chemoradiation and/or neoadjuvant and/or adjuvant immunotherapy and/or consolidation immunotherapy therapy given for locally advanced disease and developed recurrent (local or metastatic) disease ≥ 6 months of completing therapy are eligible.
* Be planned/eligible to receive first-line therapy in the advanced/metastatic setting.
* Have testing status for PDL1 tissue status.
* Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with any grade endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible.
* Adequate organ function.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 180 days after the last dose if treated with pembrolizumab plus chemotherapy, or 120 days after the last dose if treated with pembrolizumab monotherapy. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of barrier contraception starting with the first dose of study therapy through 180 days after the last dose if treated with pembrolizumab plus chemotherapy.

Cohorts 1, 2a and b: Exclusion Criteria:

* Does not plan or is ineligible to receive pembrolizumab with or without chemotherapy per institutional standard/treating provider.
* History of allogenic tissue/solid organ transplant.

Cohort 2a and b Only: Exclusion Criteria:

* Received prior treatment chemotherapy and/or immune checkpoint inhibitor therapy in the advanced/metastatic setting for lung cancer.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at doses

  ≥ 10 mg prednisone or any other form of systemic immunosuppressive therapy at C1D1. Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted (i.e., ≤ 10 mg/day prednisone equivalents). A brief course (≤ 7 days) of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Has active autoimmune disease that has required active systemic treatment in the past 2 years [i.e., with use of disease modifying agents, corticosteroids in doses greater than 10 mg of prednisone daily (or equivalent) or immunosuppressive drugs]. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, that would substantially increase the risk of incurring adverse events (AEs) from the study medications, that would interfere with the subject's participation for the full duration of the study or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has received a live vaccine within 30 days of planned start of study therapy.

Cohorts 1, 2a and b: Exclusion Criteria:

* Has received an investigational agent or has used an investigational device within 3 weeks prior to study intervention administration.
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has known untreated central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they have completed radiation therapy (where applicable), are clinically stable and have not required steroid treatment at ≥ 10 mg of prednisone for at least 3 days prior to the first dose of study intervention.
* Severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients or has a known sensitivity as applicable to carboplatin, cisplatin, taxane or pemetrexed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Real World Overall Survival (rwOS) | Up to 36 Months
  Real-world overall survival (rwOS) is defined as the length of time from the date the patient initiates treatment to the date of death or end of follow up, whichever occurred earliest.
Cohort 2 Arm A: Progression Free Survival (PFS) | Up to 36 Months
  Progression free survival is defined as the length of time from date of patient starts treatment to date of progression event or death.
Cohort 2 Arm B: Progression Free Survival (PFS) | Up to 36 Months
  Progression free survival is defined as the length of time from date of patient starts treatment to date of progression event or death.

SECONDARY OUTCOMES:
Cohort 1: Baseline ctDNA | At Baseline
  Baseline ctDNA will be summarized by mean, median, minimum, maximum, standard deviation, and coefficient of variation.
Cohort 2: Arm A and Arm B Objective Response Rate (ORR) | Up to 36 Months
  Objective response rate will be determined by summing the rates of complete response and partial response.
Cohort 2: Arm A and Arm B Overall Survival (OS) | Up to 36 Months
  Overall Survival is defined as the length of time from the date the patient initiates treatment to the date of death or end of follow up, whichever occurred earliest.

CONTACTS AND LOCATIONS:
Overall Officials: Jhanelle Gray, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland